CLINICAL TRIAL: NCT02222727
Title: Effects of Donepezil on Regional Cerebral Blood Flow Following Aneurysmal Subarachnoid Haemorrhage
Acronym: DASH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CT scanner software incompatible
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.0099; 2013-002457-30 (EudraCT Number)
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Delayed Neurological Deficit; Delayed Cerebral Ischemia; Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Active Comparator): Participants in the donepezil arm will receive the drug for 21 days as specified in the protocol in addition to current best medical treatment for aSAH patients.
  Interventions: Drug: Donepezil
- Control (No Intervention): Control group participants will not receive a placebo drug but will undergo cerebral blood flow imaging in the same manner as the donepezil patients. All other aspects of treatment will be identical to that of aSAH patients not involved in the study.

INTERVENTIONS:
Drug: Donepezil — Loading 20 mg dose of donepezil on first day of recruitment followed by once daily 5 mg dose for subsequent twenty days
  Other Names: Aricept
  Arms: Donepezil

SUMMARY:
Introduction

Aneurysmal subarachnoid hemorrhage (aSAH) is bleeding around the under surface of the brain caused by rupture of an aneurysm arising from a blood vessel. Stroke may occur in approximately one third of patients as a result of narrowing of the blood vessels around the brain, following aSAH.

One theory as to why this may happen is because bleeding around the base of the brain damages particular cells (neurons) that control blood flow around the rest of the brain. These neurons may control blood flow by releasing a neurotransmitter called Acetyl Choline (ACh). Our hypothesis is that damage to these neurons may prevent the production of ACh, which then causes reduced blood flow and stroke if left untreated.

By stimulating these neurons, we aim to investigate whether it is possible to improve the blood flow around brain and ultimately prevent strokes in patients following subarachnoid haemorrhage. Donepezil, a drug widely used in dementia, inhibits the brain's natural break down of ACh. We predict that by increasing the amount of Ach in these neurons, donepezil may improve blood flow to the brain, reducing the chance of developing stroke.

Trial Protocol

All patients admitted to St George's hospital with a confirmed aneurysmal subarachnoid haemorrhage between the ages of 18 and 85 years old will be invited to participate in the trial. The protocol has been designed to take place around the patients' aneurysm treatment, which is performed under general anesthesia (GA). Recruited participants will be anesthetized for their aneurysm treatment and then enter the study.

All trial participants will have a Xenon CT scan under GA to assess brain blood flow prior to having treatment of their aneurysm. Patients randomized to donepezil treatment will receive a loading dose of 20mg via a feeding tube immediately after their Xenon scan. Patients in the control group will not receive the drug.

All patients in the trial will undergo repeat Xenon perfusion scanning under GA between 3 and 4 hours after their first scan, which coincides with the completion of their aneurysm treatment. Those in the donepezil group will then receive a daily dose of 5 mg for a period of 21 days.

All aspects of care other than those related to the trial will be the same as for any other subarachnoid haemorrhage patients. Patients (or their legal representative for those unable to consent) will be able to decline participation in the trial or withdraw at any point.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 85 years
* Fisher score 2-4
* recruitment within 12 - 72 hours of hemorrhage

Exclusion Criteria:

* pregnancy
* breast feeding
* allergy to donepezil or other piperidine derivatives
* participants unwilling to use appropriate birth control up to 6 weeks after enrolment
* known dementia
* severe liver failure (Child-Pugh C)
* sick sinus syndrome or other supraventricular cardiac conduction abnormalities
* inspired oxygen requirement greater than 60%
* history of brittle asthma or obstructive airway disease
* aneurysm unsuitable for endovascular coiling
* concomitant use of cholinesterase inhibitor (e.g. rivastigmine, galantamine, etc)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | Within 3-4 hours of receiving drug
  Baseline xenon perfusion CT (XeCTP) scan performed immediately before donepezil loading dose administered. Follow-up XeCTP scan minimum of 3 hours after loading dose.
  For control group patients, baseline XeCTP scan performed before aneurysm treatment and follow-up scan 3-4 hours after first scan.

SECONDARY OUTCOMES:
Number of participants with adverse events. | 6 weeks from enrolment
  Participants receiving donepezil will continue to take for 21 days in total and the washout period for the drug is approximately 2 weeks accounting for a total evaluation period of 5-6 weeks.
  All participants will be regularly evaluated by clinical staff while inpatients under care of the neurosurgical service. Those discharged prior to the 6 week period will be followed up regularly by telephone and provided with a diary to record potential adverse events.
Disability assessment | 6 months from enrolment
  All participants will have a modified Rankin Score (mRS) at 6 months to assess their level of disability in comparison with their status on enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Madigan, FRCR, Study Director — St George's Hospital NHS Trust; Ramanan Sivakumaran, MRCS, Principal Investigator — St George's, University of London; Marios Papadopouos, MD FRCS(SN), Principal Investigator — St George's, University of London; Kunle Mduaoi, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, United Kingdom